CLINICAL TRIAL: NCT04608734
Title: Efficacy of Buccal Versus Intranasal Route of Administration of Midazolam Spray in Behavior Management of Pre-School Dental Patients
Brief Title: Buccal Versus Intranasal Route of Administration of Midazolam Spray in Behavior Management of Pre-School Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nourhan M.Aly (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Sponsor-Investigator, Nourhan M.Aly, Assistant Lecturer of Dental Public Health, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Buccal vs intranasal midazolam
Record Dates: First submitted 2020-10-24; First posted 2020-10-29 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Dental Anxiety

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Buccal midazolam (Experimental)
  Interventions: Drug: Buccal midazolam
- Intranasal midazolam (Active Comparator)
  Interventions: Drug: Intranasal midazolam

INTERVENTIONS:
Drug: Buccal midazolam — The drug was sprayed in the buccal vestibule across the area between the primary first and second molars in all four quadrants to maximize the absorption through wide area of the buccal mucosa.
  Arms: Buccal midazolam
Drug: Intranasal midazolam — Half of the dose was sprayed in the right nostril and the other half in the left nostril to double the absorptive surface area by short and quick puffs.
  Arms: Intranasal midazolam

SUMMARY:
Purpose of this study was to assess the efficacy of aerosolized midazolam, introduced through buccal versus intranasal mucosa in managing uncooperative children undergoing dental treatment.

DETAILED DESCRIPTION:
Thirty six children fulfilling the requirements of having a dental condition that needed treatment in two dental settings, not exceeding thirty minutes each. They were randomly assigned to one of two groups, according to the treatment offered at the first visit. At the first visit, either buccal or intranasal aerosolized midazolam was administered. At the second visit the alternate route was implemented in a cross-over design with a one week washout period. Vital signs were recorded at baseline and at 5 minutes interval throughout the treatment session.

ELIGIBILITY:
Inclusion Criteria:

* Negative and definitely negative behavior according Frankl's scale.
* ASA Group I (normal healthy patient without systemic disease) and II (patient with mild systemic disease) with no medical contraindication which rules out the use of midazolam.
* Children with at least two carious lesions requiring dental intervention in two settings of not more than 30 minute each.

Exclusion Criteria:

* Children with multiple carious lesions who require treatment under general anesthesia.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2015-06-10 (Actual); Primary Completion 2016-06-13 (Actual); Study Completion 2016-06-25 (Actual)

PRIMARY OUTCOMES:
Acceptance of drug administration | during the sedation procedure
  Assessed by a 3 point Likert scale as follows: (1) the child accepted the drug readily. 2 (fair) the child accepted the drug with some resistance. 3 (poor) the child accepted the drug with great resistance. 4 (refused) the child refused but drug administration was possible after persuasion.
Sleep score | after 5 minutes
  This will be assessed using modified Houpt scale for behavior rating:
  1. Awake, alert.
  2. Drowsy, disoriented.
  3. Intermittently asleep.
  4. Sound asleep.
Crying score | after 5 minutes
  This will be assessed using modified Houpt scale for behavior rating:
  1. Hysterical, demands attention.
  2. Continuous, making treatment difficult.
  3. Intermittent, mild, does not interfere with treatment.
  4. No crying present.
Head/oral resistance score | after 5 minutes
  This will be assessed using modified Houpt scale for behavior rating:
  1. Turns head, refuses to open mouth.
  2. Mouth closing, must request to open.
  3. Chocking, gagging, spitting.
  4. No head/oral resistance present.
Overall behavior | immediately after completion of the dental treatment procedures
  This will be assessed using modified Houpt scale for behavior rating:
  1. Aborted, no treatment performed.
  2. Very poor, treatment interrupted, partial treatment completed.
  3. Fair, difficult, all treatment completed.
  4. Good, some limited crying or movement.
  5. Excellent, no crying or movement.

CONTACTS AND LOCATIONS:
Overall Officials: Yousr N Mowafy, M.Sc, Principal Investigator — Faculty of Dentistry, Alexandria University, Egypt; Nadia A Wahba, PhD, Study Director — Faculty of Dentistry, Alexandria University, Egypt; Tamer M Ghoneim, PhD, Study Chair — Faculty of Medicine, Alexandria University, Egypt; Ghada M Mahmoud, PhD, Study Chair — Faculty of Dentistry, University of Modern Sciences and Arts, Egypt.
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt

REFERENCES:
- [Background] Chopra R, Marwaha M. Assessment of buccal aerosolized midazolam for pediatric conscious sedation. J Investig Clin Dent. 2015 Feb;6(1):40-4. doi: 10.1111/jicd.12062. Epub 2013 Dec 20. PMID 24357534
- [Background] al-Rakaf H, Bello LL, Turkustani A, Adenubi JO. Intra-nasal midazolam in conscious sedation of young paediatric dental patients. Int J Paediatr Dent. 2001 Jan;11(1):33-40. doi: 10.1046/j.1365-263x.2001.00237.x. PMID 11309871
- [Background] Kupietzky A, Houpt MI. Midazolam: a review of its use for conscious sedation of children. Pediatr Dent. 1993 Jul-Aug;15(4):237-41. No abstract available. PMID 8247896
- [Background] Kupietzky A, Holan G, Shapira J. Intranasal midazolam better at effecting amnesia after sedation than oral hydroxyzine: a pilot study. Pediatr Dent. 1996 Jan-Feb;18(1):32-4. PMID 8668567
- [Background] Primosch RE, Guelmann M. Comparison of drops versus spray administration of intranasal midazolam in two- and three-year-old children for dental sedation. Pediatr Dent. 2005 Sep-Oct;27(5):401-8. PMID 16435641
- [Background] Houpt MI, Weiss NJ, Koenigsberg SR, Desjardins PJ. Comparison of chloral hydrate with and without promethazine in the sedation of young children. Pediatr Dent. 1985 Mar;7(1):41-6. No abstract available. PMID 3857559